CLINICAL TRIAL: NCT04637880
Title: 25- Hydroxyvitamin D Levels in Pregnancy and Effects on Pregnancy Related Disorders
Acronym: VIDIS
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Ratiopharm GmbH (Industry)
Responsible Party: Principal Investigator, Julia Wild, MD, Dr. med. univ, Medical University of Vienna
Other Study IDs: V02
Record Dates: First submitted 2014-06-21; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Vitamin d Deficiency; Preeclampsia; Preterm Delivery; Gestational Hypertension; Gestational Diabetes
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia; Premature Birth; Hypertension, Pregnancy-Induced; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Evaluation of 25- Hydroxyvitamin D levels in pregnant women in Austria and potential related disorders

Hypothesis:

Austrian pregnant women are Vitamin D deficient Present vitamin D supplementation in pregnancy is insufficient Vitamin D deficiency is associated with pregnancy related disorders like preeclampsia

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* informed consent

Exclusion Criteria:

* chronic hypertension
* kidney disease
* lupus erythematodes
* diabetes mellitus
* malabsorption syndrome
* hyperparathyroidism
* surgery on the thyroid gland

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy pregnant women
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2012-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
25- Hydroxyvitamin D and relation to development of preeclampsia | over course of pregnancy

SECONDARY OUTCOMES:
25 Hydroxyvitamin D in newborn | once at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Harald Zeisler, Univ. Prof. Dr., Principal Investigator — MUV
Locations (1):
- Department of Obstetrics and fetomaternal Medicine, Medical University of Vienna, Vienna, Austria